CLINICAL TRIAL: NCT03195413
Title: Early Ultrasound-guided Nerve Block for Painful Hand Injuries in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Arvin Akhavan, Resident Physician, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001627
Record Dates: First submitted 2017-06-17; First posted 2017-06-22 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Hand Injuries; Hand Injuries and Disorders
Keywords: Hand blast injury; Nerve block; Hand injury; Forearm nerve block; Ultrasound guided nerve block; Ultrasound nerve block; Emergency department; Emergency physician; Emergency room
MeSH Terms: conditions — Hand Injuries; Disease; Emergencies | interventions — Nerve Block; Lidocaine; Epinephrine; Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nerve Block Arm (Experimental): This group of patients will receive an ultrasound-guided forearm block intervention by the study team. The nerve block will be achieved with a solution of 1% lidocaine without epinephrine and 0.5% bupivacaine without epinephrine (mixed in a 1:1 volume ratio) dosed once. A second dose will be given only in the case of complete block failure.
  Interventions: Procedure: Ultrasound-guided forearm nerve block; Drug: 1:1 volume measured solution of: 1% lidocaine without epinephrine and 0.5% bupivacaine without epinephrine; Device: Bedside ultrasound machine
- Control Arm (No Intervention): This group will receive the standard of care in our emergency department, as determined by their primary team. If a patient here receives a nerve block from the primary team, they will be handled with intention-to-treat analysis.

INTERVENTIONS:
Procedure: Ultrasound-guided forearm nerve block — An ultrasound machine will be used to identify the median, radial, and ulnar nerves in the forearm, so that a needle may be used to apply lidocaine into the soft tissue space around those nerves.
  Other Names: Nerve block
  Arms: Nerve Block Arm
Drug: 1:1 volume measured solution of: 1% lidocaine without epinephrine and 0.5% bupivacaine without epinephrine — This is the anesthetic solution that will be administered during the ultrasound-guided nerve block
  Arms: Nerve Block Arm
Device: Bedside ultrasound machine — This is the device that will be used to visualize tissues during the ultrasound-guided nerve block.
  Arms: Nerve Block Arm

SUMMARY:
This study aims to determine whether early initiation of temporary nerve block therapy improves patient satisfaction, decreases patient pain and discomfort, decreases the use of dangerous medications such as narcotics, and frees hospital resources. Hand injuries, such as blast injuries from fireworks, can be very painful. In the emergency department, providers generally use narcotic pain medications to control pain, but these have significant side effects. It is possible that temporary nerve blocks, guided by ultrasound, can be safe and useful in the emergency department. They have been shown to be effective in several studies around the country. The goal of this study is to build on the experience of others to increase the use of US-guided regional nerve blocks as a form of pain management in hand and distal forearm injuries in the Harborview Medical Center (HMC) emergency department. By working with a multidisciplinary team, the study investigators hope to use this technique to decrease narcotic use and improve pain control, and to provide important data for Emergency Medicine physicians elsewhere who are considering incorporating this nerve block technique into their practice.

DETAILED DESCRIPTION:
Hand and forearm pain secondary to fracture, laceration, dislocation, infection, and blast injury is a common issue in the emergency department (ED). Pain control is particularly important in these patients as they frequently require manipulation of their injured extremity for suturing, reduction, splinting, or abscess drainage. Pain management has traditionally centered on the use of parenteral narcotics. These medications can have significant side effects, especially in the elderly and those with comorbid diseases, and may not provide sufficient pain control in these cases, specifically in those with opioid tolerance or gruesome blast injuries. Regional nerve blocks have proven a useful tool in the management of extremity pain but have been traditionally limited to use by anesthesiologists in order to limit side effects such as intravascular infiltration and nerve damage. However, the use of direct visualization with ultrasound (US) can minimize these risks and emergency medicine (EM) physicians are using nerve blocks with increasing frequency. Recent emergency medicine literature has been promising with regard to the successful use of US-guided regional nerve blocks for finger reduction, upper extremity fractures, dislocations, abscess drainage, and hand blast injuries in the emergency department. In one case series, nerve blocks were used successfully in pediatric patients and studies measuring feasibility have found that these blocks can be done in less than ten minutes, and without significant complications. However, more studies are needed before these blocks become standard of care in all institutions. Studies that evaluate the use of other pain medications in the setting of these blocks would be particularly helpful.

Academic institutions are using US-guided nerve blocks with increasing frequency. In a recent publication 121 academic instructions provided information on usage of this technique. 84% of programs perform US-guided nerve blocks, most commonly forearm nerve blocks (ulnar, median, or radial nerves). Nerve block technique is taught via didactic sessions, online resources, and supervised training. However, most of the programs do not have specific agreements with other specialty services with regard to performing US-guided nerve blocks in the ED. One group has successfully created a multidisciplinary approach to treat blast injuries to the hand which includes EM physicians and surgeons. This team recognized the importance of surgical evaluation prior to nerve block in blast injuries to assess for risk of compartment syndrome. No cases of compartment syndrome were reported in this case series and pain control provided by the nerve block allowed the surgical team to evaluate the extent of injuries, irrigate the wound thoroughly, and employ temporizing measures such as sutures and splints while the patient waited for definitive management.

However, this aforementioned study was inherently limited in that it was a feasibility study. While promising, further work that establishes forearm blocks by ED physicians in the setting of severe hand injuries as safe and effective can guide us as to whether this mode of pain management should be standard of care. A major goal of this study will be to provide important data for emergency physicians when they consider whether or not to include these blocks into their practice.

To that end, the study investigators present a randomized controlled trial where patients with blast injuries will be randomized to standard-of-care versus early ultrasound-guided nerve block as an intervention. Measured outcomes will include pain scores, complications, and opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Patient with moderate to severe hand blast injury or other significantly painful hand or distal forearm injury Also, patients who...
* Are awake and alert
* Are able to endorse or rate their pain
* Require intravenous pain medication for their hand injury
* Are determined to be clinically sober for consent. They will need to be fluent of speech and able to articulate understanding of the procedure they will undergo and the study they will enter.

Exclusion Criteria:

Patient's who...

* Require surgical management, within one half hour, for any injury
* Require any emergent care, including resuscitation, the should preclude their regional pain management
* Are hemodynamically unstable
* Have signs of coagulopathy
* Have clinical features suggestive of compartment syndrome of the forearm, including:

  * Tense or firm forearm compartment
  * Expanding hematoma
  * Regional neurologic deficit (weakness or numbness)
* Have weakness or a sensory deficit in an intact part of their hand or forearm
* Have a vascular injury proximal to the hand
* Are unconscious or otherwise unable to endorse or rate their pain
* Are not deemed clinically sober enough to articulate an understanding of the procedure they will undergo and the study they will enter.
* Are prisoners
* Are <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-10 (Actual); Study Completion 2018-07-10 (Actual)

PRIMARY OUTCOMES:
Pain Score (1-100 visual or verbal scale) | 3 hour
  Pain score (1-100 visual or verbal scale) at 3 hours post-block

SECONDARY OUTCOMES:
Complications | 4 weeks
  Complications from the nerve blocks (i.e. compartment syndrome, persistent nerve symptoms) will be measured on follow up.
Opioid medication use | 1 day
  The amount (in morphine equivalents) number of doses of opioid medications used in the emergency department will be measured.
Additional pain scores (1-100 visual or verbal scale) | 0 - 3 hours
  Pain scores (1-100 visual or verbal scale) at time of block, 15 minutes after block, and one hour after block, and 2 hours after block.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vrablik, DO, Study Director — University of Washington Emergency Medicine
Locations (1):
- Harborview Medical Center / University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung KC, Spilson SV. The frequency and epidemiology of hand and forearm fractures in the United States. J Hand Surg Am. 2001 Sep;26(5):908-15. doi: 10.1053/jhsu.2001.26322. PMID 11561245
- [Background] Patanwala AE, Keim SM, Erstad BL. Intravenous opioids for severe acute pain in the emergency department. Ann Pharmacother. 2010 Nov;44(11):1800-9. doi: 10.1345/aph.1P438. Epub 2010 Oct 26. PMID 20978218
- [Background] Williams SR, Chouinard P, Arcand G, Harris P, Ruel M, Boudreault D, Girard F. Ultrasound guidance speeds execution and improves the quality of supraclavicular block. Anesth Analg. 2003 Nov;97(5):1518-1523. doi: 10.1213/01.ANE.0000086730.09173.CA. PMID 14570678
- [Background] Marhofer P, Greher M, Kapral S. Ultrasound guidance in regional anaesthesia. Br J Anaesth. 2005 Jan;94(1):7-17. doi: 10.1093/bja/aei002. Epub 2004 Jul 26. PMID 15277302
- [Background] Witwicki T, Dziak A. [Sarcomatous degeneration in the course of Recklinghausen's neurofibromatosis]. Chir Narzadow Ruchu Ortop Pol. 1969;34(6):809-11. No abstract available. Polish. PMID 4983335
- [Background] Stone MB, Price DD, Wang R. Ultrasound-guided supraclavicular block for the treatment of upper extremity fractures, dislocations, and abscesses in the ED. Am J Emerg Med. 2007 May;25(4):472-5. doi: 10.1016/j.ajem.2006.08.019. PMID 17499669
- [Background] Wroe P, O'Shea R, Johnson B, Hoffman R, Nagdev A. Ultrasound-guided forearm nerve blocks for hand blast injuries: case series and multidisciplinary protocol. Am J Emerg Med. 2016 Sep;34(9):1895-7. doi: 10.1016/j.ajem.2016.06.111. Epub 2016 Jul 11. No abstract available. PMID 27461885
- [Background] Frenkel O, Liebmann O, Fischer JW. Ultrasound-guided forearm nerve blocks in kids: a novel method for pain control in the treatment of hand-injured pediatric patients in the emergency department. Pediatr Emerg Care. 2015 Apr;31(4):255-9. doi: 10.1097/PEC.0000000000000398. PMID 25803747
- [Background] Liebmann O, Price D, Mills C, Gardner R, Wang R, Wilson S, Gray A. Feasibility of forearm ultrasonography-guided nerve blocks of the radial, ulnar, and median nerves for hand procedures in the emergency department. Ann Emerg Med. 2006 Nov;48(5):558-62. doi: 10.1016/j.annemergmed.2006.04.014. Epub 2006 Jun 14. PMID 17052557
- [Background] Amini R, Kartchner JZ, Nagdev A, Adhikari S. Ultrasound-Guided Nerve Blocks in Emergency Medicine Practice. J Ultrasound Med. 2016 Apr;35(4):731-6. doi: 10.7863/ultra.15.05095. Epub 2016 Mar 1. PMID 26931789